CLINICAL TRIAL: NCT05007015
Title: Transanal Irrigation for the Management of Low Anterior Resection Syndrome (LARS): A Multicenter Crossover Randomized Controlled Trial
Brief Title: Transanal Irrigation for the Management of LARS
Acronym: TAI-LARS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Assistant Professor of Surgery, McGill University, Jewish General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-05-2022-2925
Record Dates: First submitted 2021-08-10; First posted 2021-08-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer
Keywords: Transanal irrigations; Quality of Life
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled crossover trial
Masking Description: Allocation with be generated by a centralized computer generated randomized sequence to ensure allocation concealment.
  Data analyst will be blinding to treatment group but no other masking is feasible given the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transanal Irrigation (Experimental): This group will be instructed on the use of TAI to be perform daily for the three month duration of their treatment arm
  Interventions: Procedure: Transanal Irrigation
- Tradition care Control arm (No Intervention): This group tradition care group will have no modification to the care they have received prior to commencing the study. The patients in this group will use the usual dietary modifications and medications prescribed by the treating team to manage their LARS. No changes will be made to the treatment regime prescribed by their surgeon.

INTERVENTIONS:
Procedure: Transanal Irrigation — Each participant will receive a mailed package of TAI materials, given access to the LARS website, and have two scheduled virtual visits with a trained research nurse to learn how to use TAI once assigned to the intervention arm. These sessions will include one on one session with the nurse for review of the material, discussion of the device and any questions. TAI involves introducing an applicator into the anus for irrigation. An initial volume of 1000 mL will be suggested but can be increased to 1500 mL or reduced to 500 mL as per patient preference and tolerance. Applicators are single-use instruments that can be disposed of into standard waster receptacle after each treatment. The irrigation system is multiple-use and can be used for the duration recommend by the manufacturer manual. Daily irrigation can take anywhere between 20 and 90 minutes depending on individual patient experience.
  Arms: Transanal Irrigation

SUMMARY:
This study aims to evaluate the impact of Transanal irrigation (TAI) on the quality of life and low anterior resection symptoms (LARS) in Canadian rectal cancer survivors living with minor to major LARS. It proposes to teach TAI through a novel online platform and to provide virtual nursing support for the participants. To our knowledge, this is the first North American based and largest randomized control trial on the use of TAI for patients with LARS. This will also be the first study to teach and support patients through the TAI process using a virtual platform. While TAI has been demonstrated to reduce LARS scores and increased QoL in patients with significant LARS, its feasibility and acceptance for Canadian patients remains uncertain. Furthermore despite the existing studies, the rate of TAI seems to be low in North America. The hypothesis is that TAI, taught and supported through an online portal dedicated to LARS patients, will positively impact QoL and improve LARS symptoms. The results of this trial may allow TAI to become part of the standard armamentarium that clinicians offer patients for LARS management, with the presence of online nursing support and guidance to facilitate this practice.

DETAILED DESCRIPTION:
Low anterior resection syndrome (LARS) is a constellation of bowel symptoms which occur following rectal cancer treatment. These symptoms have a well characterized negative impact on a patient's quality of life (QoL) following sphincter sparing surgery. The treatment of LARS is primarily based on the management of symptoms with conservative measures such as dietary changes and fiber supplements, anti-diarrheal medications and pelvic floor physiotherapy. Despite these measures, patients often still experience uncontrolled debilitating symptoms.

Transanal irrigation (TAI) has been described for the management of LARS symptoms that persist after conservative measures have been insufficient. The positive impact of this treatment on LARS and the number of bowel movements experienced by patients has been demonstrated in several, primarily European small studies. This multicenter, assessor-blinded, parallel-group randomized control trial (RCT) will assess the outcomes of an online, nurse-led, North American TAI program for the management of LARS.

This RCT will recruit patients who have undergone a low anterior resection (LAR) with closure of any diverting stoma at least 6 months prior to entry into the trial with a LARS score of >20 at recruitment. Participants will be recruited from five academic hospitals with high volumes of rectal cancer care in Ontario and Quebec, and will be randomized using a computer-generated sequence in balanced blocks, stratified by hospital, to the intervention (TAI) or control (traditional care) arms.

Participants in the intervention arm will be asked to perform TAI every 1-2 days for a six-month period. Teaching on the use of TAI will be given through virtual sessions with an experienced research nurse and supportive material (video and animated text) on a web-based application, eLARS. This is an established online application designed to provide quality health information for patients living with LARS created by our research group. Participants in the intervention arm of this study will be given access to a restricted transanal irrigation section on this application dedicated to this RCT with detailed written instructions and educational videos on the use of TAI. Participants in the control arm of the study will have access to the general eLARS application without the section on the transanal irrigation, and no specific change in their current management routine will be required. The required sample size for this RCT, accounting for attrition, is 99 patients. It is anticipated this patient sample can be accrued from the five interested sites within a year.

The primary outcome of the study will be health-related quality of life (QoL) as measured by the European Organization for Research and Treatment of Cancer core Quality of Life questionnaire (EORTIC-QLQ-C30), with secondary outcomes including evaluation of bowel function by the LARS score, Wexner/Cleveland Clinic Fecal Incontinence Score, and bowel diary and satisfaction with TAI. Participant demographics, disease and treatment characteristics will be obtained via hospital chart review as time of recruitment. The TAI treatment effect on global QoL will be modeled using generalized estimating equations (GEE), accounting for within-subject correlations between responses at different time-points, and possible clustering of responses among participants from the same hospital.

To our knowledge, this will be the first North American trial to assess TAI acceptance and impact on quality of life for patients living with LARS. Furthermore, this will be the largest RCT to date, and the first to use a virtual platform to deliver this service for rectal cancer survivors. This study aims to provide an additional feasible and acceptable treatment option for the management of LARS symptoms refractory to our currently limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Low anterior resection by a laparoscopic, robotic, transanal total mesorectal excision, or open approach with (or without) creation of a diverting loop ileostomy for the treatment of rectal cancer, advanced adenoma or dysplasia And
* have had their ileostomy closed (if applicable) And
* completed treatment at least 6 months ago (including ileostomy closure) And
* LARS score > 20 points

Exclusion Criteria:

* Inability to provide informed consent, including fluency in English or French language
* unable to access the internet,
* presence of an ostomy,
* no active or ongoing treatment
* anastomotic stricture, sinus or any other ongoing anastomotic complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EORTC-QLQ-C30 | Monthly for the seven months of the trial
  Quality of Life change with treatment. Scale scores are calculated by averaging items within scales and transforming average scores linearly. All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems. For more details, are available in the EORTC QLQ-C30 Scoring Manual (Fayers et al., 2001)

SECONDARY OUTCOMES:
LARS Score | Monthly for the seven months of the trial
  Bowel function over the course of treatment. Scores range from 0 to 42 0-20: No LARS 21-29: Minor LARS 30-42: Major LARS
Satisfaction Survey | Monthly for the seven months of the trial
  Satisfaction survey based on LARS Consensus Definition symptoms and consequences
Bowel diaries | Will be taken in first and last 2 week periods of each treatment groups
  Standardize measure of the number of bowel movement per day

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Keane C, Fearnhead NS, Bordeianou LG, Christensen P, Basany EE, Laurberg S, Mellgren A, Messick C, Orangio GR, Verjee A, Wing K, Bissett I; LARS International Collaborative Group. International Consensus Definition of Low Anterior Resection Syndrome. Dis Colon Rectum. 2020 Mar;63(3):274-284. doi: 10.1097/DCR.0000000000001583. PMID 32032141
- [Background] Bryant CL, Lunniss PJ, Knowles CH, Thaha MA, Chan CL. Anterior resection syndrome. Lancet Oncol. 2012 Sep;13(9):e403-8. doi: 10.1016/S1470-2045(12)70236-X. PMID 22935240
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978
- [Background] Kim MJ, Park JW, Lee MA, Lim HK, Kwon YH, Ryoo SB, Park KJ, Jeong SY. Two dominant patterns of low anterior resection syndrome and their effects on patients' quality of life. Sci Rep. 2021 Feb 11;11(1):3538. doi: 10.1038/s41598-021-82149-9. PMID 33574345
- [Background] Ekkarat P, Boonpipattanapong T, Tantiphlachiva K, Sangkhathat S. Factors determining low anterior resection syndrome after rectal cancer resection: A study in Thai patients. Asian J Surg. 2016 Oct;39(4):225-31. doi: 10.1016/j.asjsur.2015.07.003. Epub 2015 Sep 2. PMID 26340884
- [Background] Battersby NJ, Juul T, Christensen P, Janjua AZ, Branagan G, Emmertsen KJ, Norton C, Hughes R, Laurberg S, Moran BJ; United Kingdom Low Anterior Resection Syndrome Study Group. Predicting the Risk of Bowel-Related Quality-of-Life Impairment After Restorative Resection for Rectal Cancer: A Multicenter Cross-Sectional Study. Dis Colon Rectum. 2016 Apr;59(4):270-80. doi: 10.1097/DCR.0000000000000552. PMID 26953985
- [Background] Sturiale A, Martellucci J, Zurli L, Vaccaro C, Brusciano L, Limongelli P, Docimo L, Valeri A. Long-term functional follow-up after anterior rectal resection for cancer. Int J Colorectal Dis. 2017 Jan;32(1):83-88. doi: 10.1007/s00384-016-2659-6. Epub 2016 Sep 30. PMID 27695976
- [Background] Iwama T, Imajo M, Yaegashi K, Mishima Y. Self washout method for defecational complaints following low anterior rectal resection. Jpn J Surg. 1989 Mar;19(2):251-3. doi: 10.1007/BF02471596. PMID 2724726
- [Background] McCutchan GM, Hughes D, Davies Z, Torkington J, Morris C, Cornish JA; LARRIS Trial Management Group. Acceptability and benefit of rectal irrigation in patients with Low Anterior Resection Syndrome: a qualitative study. Colorectal Dis. 2017 Dec 11. doi: 10.1111/codi.13985. Online ahead of print. PMID 29226518
- [Background] Rosen H, Robert-Yap J, Tentschert G, Lechner M, Roche B. Transanal irrigation improves quality of life in patients with low anterior resection syndrome. Colorectal Dis. 2011 Oct;13(10):e335-8. doi: 10.1111/j.1463-1318.2011.02692.x. PMID 21689359
- [Background] Koch SM, Rietveld MP, Govaert B, van Gemert WG, Baeten CG. Retrograde colonic irrigation for faecal incontinence after low anterior resection. Int J Colorectal Dis. 2009 Sep;24(9):1019-22. doi: 10.1007/s00384-009-0719-x. Epub 2009 May 19. PMID 19452159
- [Background] Martellucci J, Sturiale A, Bergamini C, Boni L, Cianchi F, Coratti A, Valeri A. Role of transanal irrigation in the treatment of anterior resection syndrome. Tech Coloproctol. 2018 Jul;22(7):519-527. doi: 10.1007/s10151-018-1829-7. Epub 2018 Aug 6. PMID 30083782
- [Background] Enriquez-Navascues JM, Labaka-Arteaga I, Aguirre-Allende I, Artola-Etxeberria M, Saralegui-Ansorena Y, Elorza-Echaniz G, Borda-Arrizabalaga N, Placer-Galan C. A randomized trial comparing transanal irrigation and percutaneous tibial nerve stimulation in the management of low anterior resection syndrome. Colorectal Dis. 2020 Mar;22(3):303-309. doi: 10.1111/codi.14870. Epub 2019 Oct 21. PMID 31585495
- [Background] Gosselink MP, Darby M, Zimmerman DD, Smits AA, van Kessel I, Hop WC, Briel JW, Schouten WR. Long-term follow-up of retrograde colonic irrigation for defaecation disturbances. Colorectal Dis. 2005 Jan;7(1):65-9. doi: 10.1111/j.1463-1318.2004.00696.x. PMID 15606588
- [Background] Rosen HR, Kneist W, Furst A, Kramer G, Hebenstreit J, Schiemer JF. Randomized clinical trial of prophylactic transanal irrigation versus supportive therapy to prevent symptoms of low anterior resection syndrome after rectal resection. BJS Open. 2019 Mar 18;3(4):461-465. doi: 10.1002/bjs5.50160. eCollection 2019 Aug. PMID 31388638
- [Background] Rodrigues BDS, Rodrigues FP, Buzatti KCLR, Campanati RG, Profeta da Luz MM, Gomes da Silva R, Lacerda-Filho A. Feasibility Study of Transanal Irrigation Using a Colostomy Irrigation System in Patients With Low Anterior Resection Syndrome. Dis Colon Rectum. 2022 Mar 1;65(3):413-420. doi: 10.1097/DCR.0000000000002005. PMID 33872283